CLINICAL TRIAL: NCT04990622
Title: The Effect of Diet on Parents' Mental Health in the Postnatal Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Katie Barfoot, Lecturer, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-082-KB
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Mood; Healthy; Mothers; Fathers; Parents
Keywords: mental health; postpartum; postnatal; diet; dietary intervention; flavonoids; polyphenols
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigators who process, score and analyse data will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary flavonoid group (Experimental): Participants will be encouraged to consume 2 x flavonoid-rich food items per day from the following list of flavonoid-rich foods across 2 weeks, above what they already consume each day, typically.
  * Berry fruits (~120g) e.g. blueberries, raspberries, strawberries, blackberries, blackcurrants, mixed berries
  * 2 large squares of dark chocolate (at least 70% cocoa)
  * 4-5 cups of tea (black or green) or coffee (normal or decaf varieties)
  * 1 large glass of red wine* (250ml)
  * 1 portion of leafy green vegetables such as spinach or cabbage (~70g)
  * 1 glass (250ml) of fresh orange or grapefruit juice (not from concentrate)
  Interventions: Dietary Supplement: Flavonoid-rich diet
- Control group (No Intervention): Participants will be given no instructions regarding adding food items to their diet. They will be encouraged to continue their diet as normal for 2 weeks.

INTERVENTIONS:
Dietary Supplement: Flavonoid-rich diet — Inclusion of foods rich in flavonoids.
  Other Names: Polyphenol-rich diet
  Arms: Dietary flavonoid group

SUMMARY:
Postnatal depression (PND) is a type of depression that can occur in some parents after the birth of their baby. PND has been estimated to affect 1 in 10 new parents; mothers in particular are at an increased risk of developing PND in the first year after childbirth. Symptoms of PND include a persistent feeling of sadness or low mood, a lack of enjoyment and loss of interest in the wider world, lack of energy and feeling tired all the time, difficulty bonding with your baby, withdrawing from contact with other people and problems concentrating and making decisions. Research has shown that mothers with PND have more cognitive, behavioural and interpersonal issues, and lower mood, energy and concentration than mothers without PND. Current treatments for PND include self-help resources, support from local and national organisations, psychological therapy or antidepressants with varying success rates. Further research is required to investigate accessible, cost-effective preventions or treatments for new mothers who are at risk or have been diagnosed with PND. There is also a pressing need to investigate natural alternatives to medication, especially for breastfeeding mothers who do not want to expose their infants to pharmaceuticals through breast milk.

Flavonoids are naturally occurring compounds found in high levels in foods such as berry and citrus fruits, leafy green vegetables, tea, dark chocolate and red wine. Evidence suggests that consumption of high flavonoid foods can improve health and cognitive outcomes. Prior research investigating daily dietary flavonoid intervention in a postnatal population for 2 weeks indicated significantly higher physical quality of life and significantly lower state anxiety in mothers of infants under 1 year old, at the end of the intervention. These benefits were not observed in the control group. This data shows promise for the management of mood in a key period for mothers and their babies, where risk of PND is high.

The research aim of the current study will be to further these investigations to see whether implementation of a high flavonoid diet across a 2 week period positively affects maternal mental health, specifically mood, anxiety, depressive symptoms and perceived quality of life. The study will involve recruiting mothers of infants under 6 months old to take part in an online study investigating diet and mental health. Mothers will be assigned to either a high flavonoid diet or a control condition for 2 weeks. They will complete online questionnaires (Positive and Negative Affect Scale (PANAS), Edinburgh Postnatal Depression Scale (EPDS), Postpartum-Specific Anxiety Scale (PSAS), World Health Organization Quality of Life (WHOQOL), State-Trait Anxiety Inventory (STAI) and Food Frequency Questionnaire (FFQ) at the start (day 0) and end (day 14) of the dietary intervention. In this study, a sub-sample of fathers will also be recruited to take part in the same study to assess if dietary or mood outcomes are similar or different in this population. This pilot data will inform future research of dietary interventions in new fathers.

The study does not pose ethical issues. Participants will be asked to complete non-invasive questionnaires about their mood and quality of life. For those in the high flavonoid group the change to diet will not be extreme; this group will be encouraged to include 2 items from a list of high flavonoid foods in their daily food consumption. All participants will be provided with helplines and web links upon debrief should they wish to seek further support. The helplines provided will be Samaritans UK and PANDAs Foundation. Web links to NHS, MIND and the Association for Postnatal Illness will also be listed.

DETAILED DESCRIPTION:
The study will employ a between-groups, randomised, controlled, participant-blind design. The study will primarily recruit mothers of infants under 6 months old to take part. Participants will be invited to an online study investigating diet and mental health and will be provided with an information sheet detailing what the study entails. If participants would like to take part, they will be sent a weblink to the online study. Participants will be randomly assigned to either the intervention (consumption of high flavonoid food items) or the control (no change to diet) condition. Only the experimenters will know which group participants have been assigned to to prevent participants unconsciously biasing results.

The online study will be hosted on Jisc online surveys. Once participants open the study weblink, they will be presented with the study information sheet followed by a consent form. Once participants have consented to take part, they will be asked to provide some demographic information about themselves (e.g. age, occupation, health or psychological diagnoses, any pregnancy or birth complications) and their baby (e.g. age, sex, health diagnoses, breast or bottle feeding).

Mothers will then complete PANAS-NOW, EPDS, PSAS, WHOQOL, STAI and FFQ measures. Once completed, they either will (if in high flavonoid group) or will not (if in control group) be presented with a high-flavonoid food list and instructions for food consumption over the 2 week intervention. Those presented with the high flavonoid food list will be encouraged to consume 2 high flavonoid food items per day from the list over the next 2 weeks, above what they already consume each day typically.

Both intervention and control groups will be encouraged to fill in food logs where they will write down all food consumption every day over the 2 week period.

One and a half weeks into the intervention study participants will be reminded (via email) to complete the follow up questionnaires via a weblink when convenient for them over the next few days. They will then complete the online questionnaires (PANAS-NOW, EPDS, PSAS, WHOQOL, STAI and FFQ) via the weblink at the end of the dietary intervention (day 14). Upon completion, participants will be presented with a debrief sheet explaining the aims of the study, what the study entailed and which condition they were in. Participants will also be reminded of their right to withdraw their data from the study if they wish. Helplines and support weblinks will be provided to all participants as well as encouragement for participants to contact their GP should they wish to seek support.

Alongside recruitment of postnatal mothers, fathers will also be invited to take part in the study, recruited via the mothers that consent to take part. This is so that important pilot data can be collected on a sub-sample of postnatal fathers to assess mood outcomes in this at-risk population before and after a 2 week dietary flavonoid intervention. This will follow the same methods, procedures and measures as recruited mothers.

The study aims to recruit 80 postnatal mothers. A power analysis using GPower 3.1 rendered a total sample size of 40 as appropriate to obtain a small effect (0.3) at a power of 0.95 and alpha level of 0.05. The recruitment aim will be 80 to allow for a number of participant dropouts and to allow sufficiently powered analysis between groups at baseline.

An additional aim is to recruit a sub-sample of 20 postnatal fathers alongside the main study recruiting mothers. This is to collect important pilot data to assess whether similar or different patterns or outcomes occur in a postnatal male population to inform future research into dietary intervention in men.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included if they are a biological parent (mother or father) to an infant who is between 0-6 months old.

Exclusion Criteria:

* Participants will be excluded if they have cancer, or conditions affecting the liver, heart or kidneys, due to unknown effects on flavonoid metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Mean state anxiety | 2 weeks
  Assessed using scores from the State-Trait Anxiety Inventory- State scale measure at baseline and 2 weeks. Higher scores indicate higher levels of anxiety. This questionnaire is a measure of state and trait anxiety containing 40 items in total (20 for trait; 20 for state). Only the state scale (20 items) will be used in current research to measure situational anxiety. Participants are asked to agree or disagree with anxiety-related statements on a scale of 1-4.
Mean depressive symptoms | 2 weeks
  Assessed using scores from the Edinburgh Postnatal Depression Scale at baseline and 2 weeks. Higher scores indicate higher levels of depressive symptoms. This questionnaire contains 10 items where participants rate how they have been feeling over the past 7 days on a 4-point Likert scale. The EPDS was designed for women who are pregnant or have just had a baby and has shown to be an efficient and effective way of identifying patients at risk for perinatal depression. This measure is suitable for use in new mothers and fathers.

SECONDARY OUTCOMES:
Mean quality of life | 2 weeks
  Assessed using scores from the World Health Organization Quality of Life (short form) measure at baseline and 2 weeks. Higher scores indicate higher levels of quality of life across 4 domains: physical health, psychological, social relationships and environment. It is an abbreviated version of the 100 item WHOQOL-100 and contains 24 items. The participants need to answer questions on how they feel about their quality of life on a scale from 1-5.
Mean postpartum-specific anxiety | 2 weeks
  Assessed using scores from the Postpartum-Specific Anxiety Scale for use in Global Crises measure at baseline and 2 weeks. Higher scores indicate higher levels of postpartum anxiety. This is a 12-item short form of the 51-item PSAS and has been validated for use in rapid response research at a time of global crises (during COVID-19), making it a suitable measure of anxiety in the current COVID-19 circumstances.
Mean current affect | 2 weeks
  Assessed using scores from the Positive and Negative Affect Scale at baseline and 2 weeks. This questionnaire has 20 items that describe some feelings and emotions. The participant needs to mark how much they are experiencing these feelings on a scale from 1-5. This produces scores of Positive Affect and Negative Affect; higher scores reflect higher positive or negative mood, respectively.

OTHER OUTCOMES:
General diet | 2 weeks
  Participants will complete a food frequency questionnaire at baseline and 2 weeks. This questionnaire is adapted from the EPIC-FFQ. It has a list of foods/drinks and the participant needs to state how often they consume each food/drink to assess participants' general diet.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available in Spring 2022.
Access Criteria: TBC

REFERENCES:
- [Derived] Colombage RL, Holden S, Lamport DJ, Barfoot KL. The effects of flavonoid supplementation on the mental health of postpartum parents. Front Glob Womens Health. 2024 Mar 20;5:1345353. doi: 10.3389/fgwh.2024.1345353. eCollection 2024. PMID 38577523